CLINICAL TRIAL: NCT03661723
Title: Phase II Trial of Pembrolizumab and Reirradiation in Bevacizumab Naïve and Bevacizumab Resistant Recurrent Glioblastoma
Brief Title: Pembrolizumab and Reirradiation in Bevacizumab Naïve and Bevacizumab Resistant Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, David Reardon, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-277; 3475-787 (Other: Merck)
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Glioblastoma
Keywords: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — pembrolizumab; Bevacizumab; Re-Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Pembrolizumab + Radiation (lead-in) (Experimental): * Pembrolizumab (200 mg) will initially be administered intravenously (IV) once every 3 weeks. (De-escalation dosing frequencies = once every 4 weeks and once every 6 weeks.)
  * Re-irradiation (35 Gy) will be administered to patients 5 days per week for 2 weeks
  Interventions: Drug: Pembrolizumab; Radiation: Re-irradiation
- Pembrolizumab + Bevacizumab + Radiation (lead-in) (Experimental): * Pembrolizumab (200 mg) will initially be administered intravenously (IV) once every 3 weeks. (De-escalation dosing frequencies = once every 4 weeks and once every 6 weeks.)
  * Bevacizumab (15 mg/kg) will be administered intravenously (IV) once every 3 weeks
  * Re-irradiation (35 Gy) will be administered to patients 5 days per week for 2 weeks
  Interventions: Drug: Pembrolizumab; Drug: Bevacizumab; Radiation: Re-irradiation
- Pembrolizumab + Radiation (Experimental): * Pembrolizumab (200 mg) will initially be administered intravenously (IV) once every 3 weeks
  * Re-irradiation (35 Gy) will be administered to patients 5 days per week for 2 weeks
  Interventions: Drug: Pembrolizumab; Radiation: Re-irradiation
- Pembrolizumab + Bevacizumab + Radiation (Experimental): * Pembrolizumab (200 mg) will initially be administered intravenously (IV) once every 3 weeks
  * Bevacizumab (15 mg/kg) will be administered intravenously (IV) once every 3 weeks
  * Re-irradiation (35 Gy) will be administered to patients 5 days per week for 2 weeks
  Interventions: Drug: Pembrolizumab; Drug: Bevacizumab; Radiation: Re-irradiation

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a drug (an antibody) that may treat cancer by working with the immune system
  Other Names: Keytruda
Drug: Bevacizumab — Bevacizumab (also known as "Avastin") is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.
  Other Names: Avastin
  Arms: Pembrolizumab + Bevacizumab + Radiation; Pembrolizumab + Bevacizumab + Radiation (lead-in)
Radiation: Re-irradiation — Radiotherapy destroys cancer cells using radiation aimed at a cancer from a machine

SUMMARY:
This research study is studying pembrolizumab and re-irradiation as possible treatments for glioblastoma.

The drugs involved in this study are:

* Pembrolizumab
* Radiation
* Bevacizumab, an FDA-approved drug for treating recurrent glioblastoma multiforme (GBM)

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

How the Study Interventions work:

Pembrolizumab: Pembrolizumab has been studied in lab experiments and in other types of cancer, and information from these studies suggests that it may be beneficial in this type of cancer. Pembrolizumab is a drug (an antibody) that may treat cancer by working with the immune system.

The FDA (the U.S. Food and Drug Administration) has not approved pembrolizumab for this specific disease but it has been approved for other uses.

Radiation (Re-irradiation): Radiotherapy destroys cancer cells using radiation aimed at a cancer from a machine.

The FDA (the U.S. Food and Drug Administration) has approved re-irradiation as a treatment option for this disease.

Bevacizumab: Bevacizumab (also known as "Avastin") is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.

The FDA (the U.S. Food and Drug Administration) has approved bevacizumab as a treatment option for this disease.

In this research study, the investigators are looking to determine if this combination (pembrolizumab + re-irradiation) proves helpful in treating this cancer. If the participant has already been receiving bevacizumab, the participant will continue to receive this along with pembrolizumab and re-irradiation. By doing this, the investigators will look to determine if this combination (pembrolizumab and bevacizumab + re-irradiation) proves helpful in treating this cancer.

This study will also test the safety and tolerability of this combination (pembrolizumab + re-irradiation) when given alone or with bevacizumab

ELIGIBILITY:
INCLUSION CRITERIA:

1.1 Histologically confirmed World Health Organization (WHO) Grade IV glioblastoma. Patients with original histology of low-grade glioma and subsequent histological diagnosis of GBM are eligible. Other WHO grade IV glial neoplasms such as gliosarcoma are NOT eligible 1.2 Willing and able to provide written informed consent/assent for the trial 1.3 ≥ 18 years of age on day of signing informed consent 1.4 Karnofsky performance status (KPS) ≥ 70 (Appendix A) 1.5 Unequivocal evidence for tumor progression by MRI scan 1.6 MRI within 14 days prior to start of study therapy (with vascular imaging when possible). Corticosteroid dose must be stable or decreasing for at least 5 days prior to the scan. If steroids are added or the steroid dose is increased between the date of the screening MRI scan and Day 1 dose, a new baseline scan is required 1.7 Measurable disease as per Response Assessment in Neuro-Oncology (RANO) criteria 1.8 Cohort A patients must be at their first or second relapse; Cohort B patients must have progressed on no more than one prior bevacizumab-containing regimen (may have received any # of non-bevacizumab-containing regimens). Patients who were treated with prior bevacizumab but did not progress or experienced significant toxicity, are not eligible 1.9 Previous first line therapy with at least radiotherapy utilizing standard dosing of CNS radiation - for either high-grade or low-grade glial neoplasm 1.10 The following time periods must have elapsed from projected Day 1 dose:

1. At least 3 weeks from prior surgical resection
2. At least 1 week from stereotactic biopsy
3. At least 6 months from completion of prior radiotherapy (patient may still be eligible if s/he has a new area of enhancement outside the 80% isodose line of the original radiation field)
4. At least 4 weeks from cytotoxic therapy (at least 23 days for temozolomide, and at least 6 weeks from nitrosoureas)
5. At least 1 week from cancer vaccines
6. At least 6 weeks from antibodies
7. At least 4 weeks (or 5 half-lives, whichever is shorter) from other anti-tumor therapies (not including tumor treating fields or cancer vaccines); at least 1 week from NovoTTF (Optune) or other tumor treating fields and cancer vaccines
8. Cohort B patients only: Day 1 of bevacizumab on-study must be at least 3 weeks from last dose of prior course of Avastin/bevacizumab.

1.11 All clinically significant toxic effects of prior therapy must have recovered to grade 0 or 1 or pre-treatment baseline (excluding alopecia, laboratory values listed per inclusion criteria, and lymphopenia) 1.12 Adequate organ function as defined below (screening labs performed within 14 days of treatment initiation): 1.12.1 Hematologic: Absolute neutrophil count (ANC) ≥1,500 /uL; Platelets ≥100,000 / uL; Hemoglobin ≥9 g/dL or ≥5.6 mmol/L 1.12.2 Renal: Serum creatinine ≤1.5 X institutional upper limit of normal (ULN) OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥60 mL/min for participant with creatinine levels > 1.5 X institutional ULN 1.12.3 Hepatic Serum total bilirubin ≤ 1.5 X institutional ULN OR Direct bilirubin ≤ institutional ULN for participants with total bilirubin levels > 1.5 X institutional ULN; aspartate aminotransferase (AST; SGOT) and alanine aminotransferase (ALT; SGPT) ≤ 2.5 X institutional ULN (OR ≤ 5 X institutional ULN for participants with Gilberts syndrome) 1.12.4 Coagulation: International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤1.5 X institutional ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants 1.12.5 Pulmonary: Resting baseline oxygen saturation by pulse oximetry ≥92% at rest

1.13 Negative urine or serum pregnancy within 72 hours prior to registration from any woman of child-bearing potential (WOCBP), defined as any woman physiologically capable of becoming pregnant. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

1.14 WOCBP (defined above) must agree to use a highly effective method of contraception (detailed in protocol eligibility) consistently and correctly as described below during study treatment and for 120 days after study discontinuation.

1.15 Male participants must agree to use at least one of the methods of contraception detailed in protocol eligibility starting with the first dose of study therapy through 120 days after the last dose of therapy.

EXCLUSION CRITERIA:

2.1 Recurrent tumor greater than 6 cm in maximum diameter 2.2 Currently participating or plans to participate in another study of an investigational agent or using an investigational device.

2.3 Tumor primarily localized to the brainstem or spinal cord. 2.4 Presence of multifocal tumor, diffuse leptomeningeal or extracranial disease.

NOTE: Not all instances of multifocal disease will exclude a potential patient; only patients with multifocal sites of active disease will be excluded. (e.g. A patient with a previously treated lesion that remains stable would not be excluded.)

Medical History/Conditions/Concomitant Medical Illnesses:

2.5 Diagnosis of immunodeficiency. 2.6 History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator. e.g. unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements.

2.7 History of known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhage within 12 months of start of study drug.

2.8 Evidence of intratumoral or peritumoral hemorrhage on baseline MRI scan other than those that are grade ≤ 1 and either post-operative or stable on at least 2 consecutive MRI scans.

2.9 Gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE Grade > 3 within 6 months of start of study drug.

2.10 Known additional malignancy that is progressing or requires active treatment within 1 year of start of study drug, except for those treated with surgical therapy only (e.g. basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy).

2.11 Active autoimmune disease requiring systemic treatment in the past 2 years (e.g. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg thyroxine, insulin, or physiologic corticosteroid replacement for adrenal insufficiency or pituitary/hypothalamic dysfunction, etc.) is not considered a form of systemic treatment.

2.12 History of (non-infectious) pneumonitis that required steroids or has current pneumonitis.

2.13 Active infection requiring systemic therapy. 2.14 Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

2.15 Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) and is receiving antiretroviral therapy.

2.16 Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C [e.g., hepatitis C virus (HCV) RNA (qualitative) is detected].

2.17 History of non-healing wounds or ulcers, or bone refractures within 3 months of fracture.

2.18 History of arterial thromboembolism within 12 months of start of study drug.

2.19 Clinically significant cardiovascular disease within 12 months of start of study drug, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication, percutaneous transluminal coronary angioplasty/stent.

2.20 Known history of active Bacillus Tuberculosis (TB) 2.21 Known hypersensitivity to any of the study therapy products and/or any of their excipients.

2.22 Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.

Prior Therapy:

2.23 Has received prior interstitial brachytherapy, implanted chemotherapy, stereotactic radiosurgery or therapeutics delivered by local injection or convection enhanced delivery (this exclusion applies to any locally administered therapy, including intratumoral vaccines).

2.24 Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 or with an agent directed to another stimulatory or co-stimulatory T-cell receptor (eg CTLA-4, OX-40, CD137). (These therapies target checkpoint proteins on immune cells called T-Cells.PD-1 = Programmed cell death protein 1. CTLA-4 = cytotoxic T-lymphocyte-associated protein 4. OX-40 - AKA CD134 & TNFRSF4 = Tumor necrosis factor receptor superfamily, member 4) 2.25 Has received prior Vascular endothelial growth factor (VEGF) or VEGFR inhibitor therapy such as bevacizumab, cediranib, aflibercept, vandetanib, XL-184 (Cabozantinib), sunitinib, etc. (Cohort A only)

Other Meds:

2.26 Is receiving any form of immunosuppressive therapy (e.g. chronic systemic steroid therapy exceeding dosage of 10 mg daily of prednisone equivalent) within 7 days prior to the first dose of study drug.

2.27 Has received systemic immunosuppressive treatments (aside from systemic corticosteroids as described in protocol) within six months of start of study drug (such as methotrexate, chloroquine, azathioprine, etc).

2.28 Requires treatment with high dose systemic corticosteroids defined as dexamethasone > 2 mg/day or bioequivalent for at least 3 consecutive days within 2 weeks of start of study drug.

* Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Participants are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption).
* Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents.
* A brief course of corticosteroids for prophylaxis or for treatment of non-autoimmune conditions is permitted.

2.29 Requires therapeutic anticoagulation with warfarin at baseline; patients must be off warfarin or warfarin-derivative anti-coagulants for at least 7 days prior to starting study drug. (Therapeutic or prophylactic therapy with low-molecular weight heparin is allowed.) 2.30 Has received a live vaccine within 30 days prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Reardon, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University / Herbert Irving Comprehensive Cancer Center, New York, New York
  - Hospital of the University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- COH A Safety Lead-In - Dose Level 0 (200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT); COH A Phase II @ RP2D (Dose Level 0: 200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT): * Pembrolizumab (200 mg) administered intravenously (IV) once every 3 weeks.
    o Pembrolizumab is a drug (an antibody) that may treat cancer by working with the immune system
  * Re-irradiation (35 Gy) administered 5 days per week for 2 weeks o RT destroys cancer cells using radiation aimed at a cancer from a machine
- COH B Safety Lead-In - Dose Level 0 (200 mg Pembro + 15 mg/kg Bev Every 3 Weeks + 2 Weeks of RT); COH B PhII @ RP2D (Dose Level 0: 200 mg Pembro + 15 mg/kg Bev Every 3 Weeks + 2 Weeks of RT): * Pembrolizumab (200 mg) administered intravenously (IV) once every 3 weeks.
    o Pembrolizumab is a drug (an antibody) that may treat cancer by working with the immune system
  * Bevacizumab or biosimilar (15 mg/kg) administered intravenously (IV) once every 3 weeks
    o Bevacizumab is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.
  * Re-irradiation (35 Gy) administered 5 days per week for 2 weeks o RT destroys cancer cells using radiation aimed at a cancer from a machine
Period: Overall Study
Arm/Group | COH A Safety Lead-In - Dose Level 0 (200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT) | COH A Phase II @ RP2D (Dose Level 0: 200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT) | COH B Safety Lead-In - Dose Level 0 (200 mg Pembro + 15 mg/kg Bev Every 3 Weeks + 2 Weeks of RT) | COH B PhII @ RP2D (Dose Level 0: 200 mg Pembro + 15 mg/kg Bev Every 3 Weeks + 2 Weeks of RT)
Started | 6 | 24 | 6 | 24
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 24 | 6 | 24
Not completed — Disease Progression | 4 | 24 | 4 | 19
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 4
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Clinical Deterioration | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Populations are defined by treatment assignment; Safety Lead-in and Phase II patient information is reported together
Groups:
- COH A - Dose Level 0 (200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT): Inclusive of both Safety Lead-In & PH II COH A participants, as they were all treated at the same dose:
  * Pembrolizumab (200 mg) administered intravenously (IV) once every 3 weeks.
  * Re-irradiation (35 Gy) administered 5 days per week for 2 weeks
- COH B - Dose Level 0 (200 mg Pembro + 15 mg/kg Bev Once Every 3 Weeks + 2 Weeks of RT): Inclusive of both Safety Lead-In & PH II COH B participants, as they were all treated at the same dose:
  * Pembrolizumab (200 mg) administered intravenously (IV) once every 3 weeks.
  * Bevacizumab or biosimilar (15 mg/kg) administered intravenously (IV) once every 3 weeks
  * Re-irradiation (35 Gy) administered 5 days per week for 2 weeks
- Total: Total of all reporting groups
Arm/Group | COH A - Dose Level 0 (200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT) | COH B - Dose Level 0 (200 mg Pembro + 15 mg/kg Bev Once Every 3 Weeks + 2 Weeks of RT) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 22 | 48
  >=65 years | 4 | 8 | 12
Age, Continuous [Median (Full Range); unit: years] | 61 [20 to 76] | 61 [34 to 75] | 61 [20 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 16 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 26 | 17 | 43
  Unknown or Not Reported | 3 | 8 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 27 | 18 | 45
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 1 | 7 | 8
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Karnofsky performance status (KPS) [Count of Participants; unit: Participants] — Karnofsky Performance Scale (KPS):
  100 Normal, no complaints, no evidence of dz 90 Able to carry on normal activity; minor signs/symptoms of dz 80 Normal activity w effort; some signs/symptoms of dz 70 Cares for self, unable to carry on normal activity/do active work 60 Requires occasional assistance, but able to care for most needs 50 Requires considerable assistance & frequent medical care 40 Disabled; requires special care & assistance 30 Severely disabled; hospitalization indicated 20 Very sick; hospitalization indicated 10 Moribund; fatal processes progressing rapidly 0 Dead
  Participants
    KPS = 70 | 5 | 9 | 14
    KPS = 80 | 10 | 12 | 22
    KPS = 90 | 14 | 8 | 22
    KPS = 100 | 1 | 1 | 2
Current Recurrence # [Count of Participants; unit: Participants]
  First Relapse | 19 | 10 | 29
  Second Relapse | 11 | 12 | 23
  Third Relapse | 0 | 5 | 5
  Fourth Relapse | 0 | 3 | 3
Extent of Resection Prior to Study Enrollment [Count of Participants; unit: Participants]
  Gross Total Resection (GTR) | 8 | 1 | 9
  Sub-Total Resection (STR) | 6 | 0 | 6
  Biopsy | 1 | 0 | 1
  None | 11 | 29 | 40
  Unknown | 4 | 0 | 4
MGMT Methylation Status [Count of Participants; unit: Participants] — The DNA repair enzyme O(6)-methylguanine-DNA methyltransferase (MGMT) antagonizes the genotoxic effects of alkylating agents. MGMT promoter methylation is the key mechanism of MGMT gene silencing and predicts a favorable outcome in patients with glioblastoma who are exposed to alkylating agent chemotherapy.
  Participants
    Methylated | 7 | 11 | 18
    Unmethylated | 11 | 14 | 25
    Unknown | 12 | 5 | 17
IDH mutation [Count of Participants; unit: Participants]
  Present | 2 | 3 | 5
  Absent | 17 | 26 | 43
  Unknown | 11 | 1 | 12
Dexamethasone Use @ Time On Study [Count of Participants; unit: Participants]
  Receiving Dexamethasone | 6 | 13 | 19
  No Dexamethasone | 24 | 17 | 41
Time from Original GBM Diagnosis to Trial Registration [Median (Full Range); unit: months] | 13.5 [1 to 48] | 14.5 [0 to 63] | 14 [0 to 63]

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Per Response Assessment in Neuro-Oncology (RANO) Criteria:
  * Complete Response (CR):
    * Disappearance of all enhancing measurable & non-measurable disease sustained for at least 4 weeks
    * No new lesions
    * Stable or improved non-enhancing (T2/FLAIR) lesions
    * No corticosteroids (or physiologic replacement doses only)
    * And stable or improved clinically
  * Partial Response (PR):
    * >=50% decrease compared with baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks;
    * No progression of non-measurable disease
    * No new lesions
    * Stable or improved non-enhancing (T2/FLAIR) lesions
    * Same or lower dose of corticosteroids compared with baseline scan
    * And stable or improved clinically
  Overall Response Rate (ORR) = Frequency of CR + PR within a population.
Time Frame: 2 years
Population: # of participants in the analysis population who achieve a complete response (CR) or partial response (PR) using RANO criteria
Measure: Count of Participants; unit: Participants
Arm/Group | COH A - Dose Level 0 (200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT) | COH B - Dose Level 0 (200 mg Pembro + 15 mg/kg Bev Once Every 3 Weeks + 2 Weeks of RT)
Number analyzed (Participants) | 30 | 30
Participants | 1 | 3

2. Primary Outcome: Overall Survival Rate at 6 Months (OS-6)
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | COH A - Dose Level 0 (200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT) | COH B - Dose Level 0 (200 mg Pembro + 15 mg/kg Bev Once Every 3 Weeks + 2 Weeks of RT)
Number analyzed (Participants) | 30 | 30
percentage of participants | 83.3 [6.5 to 92.7] | 56.7 [37.3 to 72.1]

3. Primary Outcome: Overall Survival Rate at 12 Months (OS-12)
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | COH A - Dose Level 0 (200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT) | COH B - Dose Level 0 (200 mg Pembro + 15 mg/kg Bev Once Every 3 Weeks + 2 Weeks of RT)
Number analyzed (Participants) | 30 | 30
percentage of participants | 40.0 [22.8 to 56.6] | 16.6 [6.0 to 31.7]

4. Secondary Outcome: Safety & Tolerability: SAEs Experienced by Participants
Description: Number of Participants who Experienced an SAE Deemed At Least Possibly Related to Study Treatment (XRT, pembrolizumab, &/or bevacizumab)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | COH A - Dose Level 0 (200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT) | COH B - Dose Level 0 (200 mg Pembro + 15 mg/kg Bev Once Every 3 Weeks + 2 Weeks of RT)
Number analyzed (Participants) | 30 | 30
Participants | 6 | 7

5. Secondary Outcome: Duration of Response
Description: Each patient's response data is reviewed and the duration of his/her best response determined (in days).
Time Frame: 1 year
Population: 5 COH B patients were censored for duration of response, as they each withdrew consent to be followed (or initiated a new therapy regimen) right after a scan that showed stable disease.
Measure: Median (Full Range); unit: days
Arm/Group | COH A - Dose Level 0 (200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT) | COH B - Dose Level 0 (200 mg Pembro + 15 mg/kg Bev Once Every 3 Weeks + 2 Weeks of RT)
Number analyzed (Participants) | 30 | 25
days | 79.5 [0 to 266] | 42.0 [0 to 168]

6. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Progression is defined using Radiologic Assessment in Neuro-Oncology (RANO) criteria, as any of the following:
  * ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions compared with the smallest tumor measurement, on stable or increasing doses of corticosteroids
  * Any new enhancing measurable lesion
  * Clear clinical deterioration not attributable to other causes apart from the tumor or changes in corticosteroid dose
  * Cohort B: Significant increase in T2/FLAIR non-enhancing lesions on stable or increasing doses of corticosteroids not felt to be caused by co-morbid events
  * Clear progression of non-measurable disease
  * Or failure to return for evaluation as a result of death or deteriorating condition
Time Frame: 2 years
Measure: Median (Standard Error); unit: months
Arm/Group | COH A - Dose Level 0 (200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT) | COH B - Dose Level 0 (200 mg Pembro + 15 mg/kg Bev Once Every 3 Weeks + 2 Weeks of RT)
Number analyzed (Participants) | 30 | 30
months | 4.2 (0.4551) | 4.0 (0.5467)

7. Secondary Outcome: 6-month Progression Free Survival (PFS-6)
Description: as for outcome 6
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | COH A - Dose Level 0 (200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT) | COH B - Dose Level 0 (200 mg Pembro + 15 mg/kg Bev Once Every 3 Weeks + 2 Weeks of RT)
Number analyzed (Participants) | 30 | 30
percentage of participants | 13.3 [4.2 to 27.7] | 10.6 [2.2 to 27.0]

8. Secondary Outcome: Median Overall Survival (OS)
Time Frame: Participants were followed for survival until death; survival was followed for a max of 4 years. Other Adverse Events (AEs) were collected from registration through 30 days after last dose (SAEs through 90 days); AEs were followed for a max of 2 years.
Measure: Median (Standard Error); unit: months
Arm/Group | COH A - Dose Level 0 (200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT) | COH B - Dose Level 0 (200 mg Pembro + 15 mg/kg Bev Once Every 3 Weeks + 2 Weeks of RT)
Number analyzed (Participants) | 30 | 30
months | 11.8 (1.0262) | 8.6 (1.1766)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from registration through 30 days after last dose. Serious AEs (SAEs) were collected through 90 days after last dose (or 30 days if pt initiated new anticancer therapy). AEs were followed for a max of 2 years on this trial. Participants were followed every 3 months (+/- 1 month) until death for survival. Survival was followed for a max of 4 years on this trial.
Description: An AE is any undesirable sign, symptom or medical condition that develops or worsens in severity after initiating study treatment or any protocol-specified procedure, regardless of attribution. An SAE is any AE at any dose & regardless of causality that: results in death, is life-threatening, requires or prolongs inpatient hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly or birth defect, or is an important medical event
Arm/Group | COH A - Dose Level 0 (200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT) | COH B - Dose Level 0 (200 mg Pembro + 15 mg/kg Bev Once Every 3 Weeks + 2 Weeks of RT)
All-Cause Mortality (participants affected / at risk) | 30/30 | 28/30
Serious Adverse Events (participants affected / at risk) | 14/30 | 11/30
Other Adverse Events (participants affected / at risk) | 30/30 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | COH A - Dose Level 0 (200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT) (N=30) | COH B - Dose Level 0 (200 mg Pembro + 15 mg/kg Bev Once Every 3 Weeks + 2 Weeks of RT) (N=30)
Papilledema (Eye disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 2 | 0
Dysarthria (Nervous system disorders) | 2 | 0
Dysphasia (Nervous system disorders) | 1 | 1
Edema cerebral (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 4 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 1 | 2
Stroke (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specify: Left facial droop (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 2 | 2
Surgical and medical procedures - Other, specify: Craniotomy revision with hardware removal (Surgical and medical procedures) | 1 | 0
Surgical and medical procedures - Other, specify: Craniotomy for tumor resection (Surgical and medical procedures) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | COH A - Dose Level 0 (200 mg Pembro Once Every 3 Weeks + 2 Weeks of RT) (N=30) | COH B - Dose Level 0 (200 mg Pembro + 15 mg/kg Bev Once Every 3 Weeks + 2 Weeks of RT) (N=30)
Hyperthyroidism (Endocrine disorders) | 2 | 0
Nausea (Endocrine disorders) | 2 | 0
Fatigue (General disorders) | 12 | 4
Flu like symptoms (General disorders) | 2 | 0
Gait disturbance (General disorders) | 2 | 5
Sinusitis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 2 | 0
Upper respiratory infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 2
Fall (Injury, poisoning and procedural complications) | 3 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2
Lymphocyte count decreased (Investigations) | 7 | 3
Weight gain (Investigations) | 3 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 4
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 5 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 3 | 3
Cognitive disturbance (Nervous system disorders) | 0 | 2
Dysphasia (Nervous system disorders) | 8 | 5
Headache (Nervous system disorders) | 10 | 5
Memory impairment (Nervous system disorders) | 3 | 2
Seizure (Nervous system disorders) | 2 | 0
Agitation (Psychiatric disorders) | 2 | 2
Confusion (Psychiatric disorders) | 4 | 0
Proteinuria (Renal and urinary disorders) | 0 | 8
Urinary incontinence (Renal and urinary disorders) | 2 | 3
Hypertension (Vascular disorders) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT03661723/Prot_SAP_000.pdf